CLINICAL TRIAL: NCT07096869
Title: A Randomized, Open-Label, Two-Period, Crossover Bioequivalence Study of Paclitaxel Protein-bound Particles for Injectable Suspension (Albumin-bound) and Abraxane® in Breast Cancer Patients
Brief Title: Bioequivalence Study of Paclitaxel Protein-bound Particles for Injectable Suspension (Albumin-bound) in Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HF112-001
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel protein-bound particles for injectable suspension (albumin-bound) (Experimental): The subjects randomly reveived single dose of 260 mg/m^2 of paclitaxel protein-bound particles for injectable suspension (albumin-bound)
  Interventions: Drug: Paclitaxel protein-bound particles for injectable suspension (albumin-bound)
- Abraxane® (Experimental): The subjects randomly reveived single dose of 260 mg/m^2 of Abraxane®
  Interventions: Drug: Abraxane®

INTERVENTIONS:
Drug: Paclitaxel protein-bound particles for injectable suspension (albumin-bound) — IV infusion, 260 mg/m^2
  Arms: Paclitaxel protein-bound particles for injectable suspension (albumin-bound)
Drug: Abraxane® — IV infusion, 260 mg/m^2
  Arms: Abraxane®

SUMMARY:
The main purpose of this study is to evaluate the bioequivalence of paclitaxel protein-bound particles for injectable suspension (albumin-bound) (100 mg, test product) and Abraxane® (100 mg, reference product) in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects fully understand the purpose, nature, method and possible adverse reactions of the study, volunteer as subjects, and sign informed consent prior to the commencement of any study procedure;
* 2) Male and female, ages 18-75 years both inclusive;
* 3) Subjects with breast cancer confirmed by histopathology and/or cytology who meet one of the following conditions: ①Metastatic breast cancer, after failure of combination chemotherapy for metastatic disease or relapse within 6 months of adjuvant chemotherapy. Prior therapy should have included an anthracycline unless clinically contraindicated; ②This treatment criteria (NCCN guidelines and CSCO guidelines - Breast cancer) is used to determine whether the subjects are suitable for paclitaxel for injection (albumin-bound) monotherapy. ③Subjects received standard treatment without conditions and were judged to benefit from injectable paclitaxel (albumin-binding) monotherapy;
* 4) ECOG Score ≤ 2 points;
* 5) The expecting life span ≥ 3months;
* 6) The results of blood, liver and kidney function tests are within the following ranges: Absolute neutrophil counts (ANC) ≥ 1.5×10^9/L Platelets (PLT) ≥ 100×10^9/L Hemoglobin (Hb) ≥ 90 g/L Total bilirubin (TBIL) ≤ 1.5×ULN Alanine transaminase (ALT), Aspartate aminotransferase (AST)≤×ULN (for patients with liver metastasis, ≤ 5×ULN) Creatinine clearance (CrCL)≥ 60 mL/min
* 7) The subject has no fertility plan (including sperm donation and egg donation) for at least 6 months from the signing of informed consent to the last dose and voluntarily takes non-drug effective contraceptive measures;
* 8) Subjects can communicate well with the investigators, understand and comply with the requirements of the study.

Exclusion Criteria:

* 1) A severe allergy or hypersensitivity to paclitaxel or human albumin;
* 2) In addition to cancer, have any other serious liver, kidney/genitourinary, gastrointestinal (e.g., abdominal inflammation), cardiovascular (e.g., congestive heart failure, ventricular arrhythmia, myocardial infarction, unstable angina), cerebrovascular, pulmonary (e.g., interstitial lung disease), endocrine, immune, musculoskeletal, neurological, psychiatric, skin, or blood (e.g., bleeding diathymia or clotting disorders) diseases Patients with a known or present history of the disease who are deemed unsuitable for enrollment by the investigators;
* 3) Those who had undergone major surgery within 4 weeks prior to screening, or planned to undergo major surgery during the study period;
* 4) Pregnant or lactating female subjects;
* 5) Hepatitis B surface antigen positive and HBV DNA positive; HCV core antibody positive and HCV RNA positive; HIV antigen/antibody positive; treponema pallidum antibody positive and rapid plasma reaction hormone (RPR) positive;
* 6) Those who used chemical small molecule anti-tumor drugs (including endocrine therapy), biological macromolecular anti-tumor drugs, biological therapy, radiotherapy or needed to combine other anti-tumor drugs for treatment during the study period within 4 weeks before the first dose;
* 7) Electrocardiogram shows significant abnormality, and/or baseline QTcF interval is > 470 ms;
* 8) Pre-screening sensory neuropathy/peripheral neuropathy are ≥ grade 2;
* 9) Blood donation or significant blood loss (> 400 mL) within 90 days before - screening;
* 10) Ingestion of an inhibitor or inducer of CYP2C8 or CYP3A4 within 28 days prior to dosing (acceptable drug use is stable in homeostasis, that is, the dosing regimen remains unchanged; However, the use of moderate-strong inhibitory agents/moderate-strong inducers should be prohibited), or drugs (including Chinese herbs) that can affect the absorption, distribution, metabolism and excretion behavior of the study drugs or special diets (such as products containing caffeine or xanthine, grapefruit fruits and products containing grapefruit ingredients, etc.);
* 11) Those who consumed more than 14 units of alcohol per week in the 3 months before screening (1 unit ≈ 360 mL for beer, or 45 mL for spirits, or 150 mL for wine) or who could not stop drinking during the study period or who are breath-positive for alcohol;
* 12) Smoking > 5 cigarettes per day within 3 months prior to screening or smoking cannot be stopped during the study period;
* 13) Any clinically significant abnormal results in the subjects' vital signs, physical examination, clinical laboratory examination (unless otherwise specified in the protocol), 12-lead electrocardiogram (ECG) and other examination results that the investigator deems unsuitable for enrollment;
* 14) Within 6 months prior to screening, there is a history of drug abuse (except regular use of pain medications due to cancer pain) or positive drug abuse screening;
* 15) Toxicity caused by using of anti-tumor drugs prior to enrolment do not return to ≤ grade 1 or baseline levels, except for alopecia;
* 16) Subjects receiving granulocyte-stimulating growth factor treatment within 2 weeks before dosing;
* 17) Subjects who have participated in any clinical trial within 1 month before screening (start from the time of the last dose);
* 18) Any other circumstances determined by the investigator to be inappropriate are not suitable for participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 72 hours
  Evaluation of Peak Plasma Concentration (Cmax) of total and unbound paclitaxel
Area under the plasma concentration versus time curve AUC0-t | 72 hours
  Evaluation of Area under the plasma concentration versus time curve AUC0-t of total and unbound paclitaxel
Area under the plasma concentration versus time curve AUC0-∞ | 72 hours
  Evaluation of Area under the plasma concentration versus time curve AUC0-∞ of total and unbound paclitaxel

SECONDARY OUTCOMES:
Time to peak Plasma Concentration (Tmax) | 72 hours
  The Tmax of total and unbound paclitaxel
Elimination of half-life (t1/2) | 72 hours
  The t1/2of total and unbound paclitaxel
Incidence of Adverse Events | Up to 6 mouths
  Collection of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China